CLINICAL TRIAL: NCT02939157
Title: Pocket-sized Ultrasound for Point-of-care Diagnosis of Heart Failure
Acronym: POCUS
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-02514
Record Dates: First submitted 2016-09-20; First posted 2016-10-19 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2016-09

CONDITIONS: Heart Failure, Congestive; Cardiac Failure
Keywords: Diagnostic Ultrasound; Primary Care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cardiac diagnostic ultrasound — Point-of-care ultrasound for diagnosing heart failure in primary care patients
  Other Names: Point-of-care ultrasound

SUMMARY:
Assessment of pocket sized ultrasound (Vscan GE Healthcare) for diagnosing heart failure in primary care patients, with a comprehensive cardiac ultrasound examination (Siemens Acusan P10) performed at a specialized the eco.lab, as reference.

DETAILED DESCRIPTION:
Waiting times for cardiac ultrasound is a cause of delay in identification of heart failure, which means delayed treatment, or that treatment recommendations are based on insufficient knowledge. Heart failure is a common condition; about 10% of 80-year-old people are affected and most patients are treated within primary care. A new ultrasound technology with integrated software support for interpretation (pocket-sized ultrasound) promises to improve care for heart patients and lead to earlier treatment with effective drugs. In cooperation with Norwegian researchers and the Region of Jämtland Härjedalen, this project opens opportunities for a significant medical innovation. The new concept, pocket-sized ultrasound for diagnosis of heart failure, has not previously been validated in patients seen in primary care. A new study may provide very important information that is directly applicable in the care of heart failure patients. We aim to recruit 250 study patients from the waiting list of patients referred from GPs, to ultrasound at the dpt. Of Clinical Physiology, Östersund Hospital, due to a suspicion of heart failure. The examinations will be carried out during the same day, with the investigators blinded to each other. The new concept of ultrasound has a potential to provide more cost-effective identification and monitoring of patients with heart failure in primary care.

ELIGIBILITY:
Inclusion Criteria: Study patients fulfil all of the following criteria:

1. Age 20 and over
2. Recruited from primary care clinics, in the Region of Jämtland Härjedalen, Sweden.
3. Referred to comprehensive cardiac ultrasound (reference method) from GPs, due to suspected heart failure.
4. Provide written informed consent before enrolment.

Exclusion Criteria:

1. Non consenting patients.
2. Patients in need of acute medical attention.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250 adult study patients consulting to GPs in primary care for suspected cardiac failure.
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Cardiac failure | Assessment of cardiac failure by the study method (pocket sized ultrasound) is made on the same day as the reference method (comprehensive cardiac ultrasound), by independent investigators.
  Detection of cardiac failure in patients consulting in primary care by a pocket sized ultrasound device, for use in primary care

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Nilsson, MD;PhD, Principal Investigator — Umeå University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson G, Soderstrom L, Alverlind K, Samuelsson E, Mooe T. Hand-held cardiac ultrasound examinations performed in primary care patients by nonexperts to identify reduced ejection fraction. BMC Med Educ. 2019 Jul 25;19(1):282. doi: 10.1186/s12909-019-1713-9. PMID 31345207